CLINICAL TRIAL: NCT06499324
Title: Surgical Treatment of Large Incisional Hernia with Botulinum Toxin a Injection: a Double-blind Randomized Controlled Trial
Brief Title: Surgery with Botulinum Toxin a for Incisional Hernia
Acronym: INCISOX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220805
Record Dates: First submitted 2024-05-31; First posted 2024-07-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Incisional Hernia
Keywords: Incisional Hernia; Botulinum toxin A; Incisional Hernia repair; Laparatomy
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The injection physician and surgeon will be blinded to the randomization group due to the transparency of BTA and the placebo.
  The surgeon will not know the patient's treatment during surgery as BTA does not affect muscle appearance.
  A blinded CT-scan, four to six weeks post-injection, will be performed; results will be kept from the surgeon to avoid unblinding, and patients will remain blinded to their randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BTA group (Experimental): This arm corresponds to patients presenting with midline anterior primary or recurrent IH (subxiphoidal to suprapubic) of width >= 10 cm, without loss of domain, scheduled for IH repair with mesh.
  Patients will be injected with 288 IU of BTA (XEOMIN® 100U) into the lateral muscles (18 injection sites, 16UI/8mL/injection site), 4 to 6 weeks before the treatment of the IH.
  Interventions: Drug: BTA group
- Placebo group (Placebo Comparator): This arm corresponds to patients presenting with midline anterior primary or recurrent IH (subxiphoidal to suprapubic) of width >= 10 cm, without loss of domain, scheduled for IH repair with mesh.
  Patients will be injected with placebo of BTA (XEOMIN® 100U matching placebo) into the lateral muscles (18 injection sites, 8mL/injection site), 4 to 6 weeks before the treatment of the IH.
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: BTA group — It consists of a blind injection of 288 IU (/144mL) of BTA (XEOMIN®) into the lateral muscles (18 injection sites, 16UI/8mL/injection site), 4 to 6 weeks before the treatment of a large anterior IH (width ≥ 10 cm) with open non absorbable mesh repair. The injection of BTA (XEOMIN®) will be done during an outpatient hospitalization, in each of the 3 lateral muscles of the abdomen on each side. To do this in the BTA group, 3 vials of 100 equivalent IU of BTA (XEOMIN® 100U), diluted to 2 IU/mL with 0.9% saline will be distributed in 3 syringes of 50 mL equipped with a 21G needle. A total of 72 mL of BTA solution (144 IU) will be injected on each side, at 3 injection points between the costal rim and iliac crest, under ultrasound control.
  Arms: BTA group
Drug: Placebo group — It consists of a blind injection of placebo of BTA (XEOMIN® 100U matching placebo) into the lateral muscles (18 injection sites, 8mL/injection site), 4 to 6 weeks before the treatment of a large IH (width >= 10 cm) with open non absorbable mesh repair. The injection of placebo of BTA (XEOMIN® 100U matching placebo) will be done during an outpatient hospitalization, in each of the 3 lateral muscles of the abdomen on each side. To do this in the control group, 3 vials of placebo of BTA (XEOMIN® 100U matching placebo), diluted with 0.9% saline will be distributed in 3 syringes of 50 mL equipped with a 21G needle. A total of 72 mL of placebo of BTA solution will be injected on each side, at 3 injection points between the costal rim and iliac crest, under ultrasound control.
  Arms: Placebo group

SUMMARY:
After laparotomy, treating large incisional hernias (width >= 10cm) proves challenging due to the progressive retraction of lateral abdominal muscles and the separation of rectus muscles. This width is a significant risk factor for repair failure and recurrence. High rates of severe postoperative morbidity, up to 50%, are reported, linked to dissection extent, increased muscular tension, and abdominal pressure. Reconstructing normal anatomy by bringing muscles together may be impossible, leading to the use of complex procedures like component separation techniques (CST), involving large aponeurotomy for muscle relaxation. Intramuscular injection of botulinum toxin A (BTA) induces reversible flaccid paralysis, with potential benefits in hernia closure, known as "chemical CST." Retrospective studies suggest reduced muscle retraction and facilitated closure without specific morbidity. Prehabilitation with BTA aims to reduce surgical morbidity compared to repair and CST. The prospective evaluation of BTA's clinical benefits, including reduced postoperative morbidity, pain, successful abdominal closure, and decreased IH recurrence risk, is lacking. A prospective randomized double-blind placebo-controlled trial is proposed to demonstrate BTA's efficacy. The hypothesis is that BTA injection before IH repair is more effective than a placebo in reducing postoperative morbimortality. Secondary expectations include a significant reduction in complete closure of the abdominal wall without CST.

DETAILED DESCRIPTION:
Almost 20% of patients will develop an incisional hernia (IH) after laparotomy. Each year in France, around 30,000 patients undergo IH repair with mesh [PMSI, 2017]. The treatment of large IH (width>=10cm) is difficult due to the progressive retraction of the lateral abdominal muscles associated with the separation of the rectus muscles. The IH width is a major risk factor of failure of the repair and recurrence. Furthermore, high rates of severe postoperative morbidity, up to 50%, have been reported and related to the extent of dissection and increase of muscular tension and abdominal pressure. Thus, bringing the muscles together to reconstruct the normal anatomy may be impossible and lead the surgeon to use complex and morbid technical procedures, such as component separation techniques (CST), consisting in large aponeurotomy for relaxation of the lateral muscles. The intramuscular injection of botulinum toxin A (BTA) makes it possible to obtain a reversible flaccid paralysis of the striated muscle fibers and its advantage has been demonstrated for the treatment of neurological spasticity. Its use to obtain a relaxation of the lateral muscles of the abdomen, so-called "chemical CST", reduce their retraction and facilitate hernia closure, as studied in retrospective studies, without specific morbidity. In particular, prehabilitation with BTA injection, is supposed to reduce surgical morbidity in comparison with surgical repair and CST. The expected clinical benefit, in terms of reduction of postoperative morbidity and pain, successful closure of the abdomen, and reduction of the risk of recurrence of the IH, has never been evaluated prospectively. Thus, a prospective randomized double-blind placebo-controlled trial would be the best method to demonstrate the benefit of BTA injection. The investigators hypothesize that BTA injection in the lateral muscles before IH repair is more effective than placebo injection in reducing postoperative morbimortality. Secondarily, the investigators expect that BTA injection is associated with a significant reduction of complete closure of the abdominal wall without CST.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 79 years;
2. BMI < 35 kg/m²;
3. Midline anterior primary or recurrent IH (subxiphoidal to suprapubic), of width >= 10 cm, on the abdominopelvic CT without injection of contrast agent, performed in the 6 months before inclusion (EHS W3);
4. IH without loss of domain, defined by the ratio: (volume of the peritoneal sac) / (total peritoneal volume) < 25%, on the abdominal CT without injection of contrast agent, performed in the 6 months before inclusion;
5. Written informed consent;
6. Scheduled surgery for an open IH repair;
7. For female of childbearing potential: using highly effective contraception.

Exclusion Criteria:

1. Other types of IH (lateral, groin, para-stomal, portsite);
2. VHWG grades 3 or 4 for the risk of surgical site infection;
3. Ongoing skin infection or inflammation at the IH site or at the BTA injection site;
4. Planned IH repair with slowly absorbable mesh;
5. IH with loss of domain (volumetric ratio > 25%);
6. Emergency IH surgery;
7. ASA score > 3;
8. Pregnancy or breastfeeding;
9. Ongoing treatment with aminoglycosides;
10. Severe hemostasis disorder or non-weaning treatment with curative dose anticoagulant;
11. Active tobacco use (or cessation inferior to 3 months);
12. Use of another investigational product within 6 months or 5 half-lives (whichever is longer), or currently participating in a prospective study with an investigational product, whether it concerns an experimental drug or a medical device;
13. Patient not covered by social insurance;
14. Patient under legal guardianship;
15. Hypersensitivity to the active substance (Clostridium Botulinum neurotoxin type A) or to any of the excipients (Human albumin, sucrose);
16. Generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert-Eaton syndrome, peripheral motor neuropathic diseases (e.g. amyotrophic lateral sclerosis or motor neuropathy), facial nerve disorders, underlying neurological disorders) and history of dysphagia and aspiration);
17. Patient with ongoing treatment with medicinal products that interfere with the transfer of an impulse from a nerve to a muscle, e.g. tubocurarine-type muscle relaxants that weaken the muscles;
18. Patient with severe and uncontrolled cardiovascular diseases;
19. Patient has received BTA within 12 weeks;
20. Patients with a history of seizures.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2028-08-04 (Estimated); Study Completion 2029-03-04 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the efficacy of preoperative BTA injection in the lateral abdominal wall muscles reduces the rate of postoperative morbimortality after large IH (width >= 10cm) repair with mesh, compared with placebo injection. | During the 90-day postoperative period
  Occurrence of Clavien-Dindo classification grade II or higher post-operative complication

SECONDARY OUTCOMES:
Assessment of the impact of preoperative BTA injection on length of stay. | From surgery until hospital discharge, average 5 days
  Length of hospital stay in days
Assessment of the impact of preoperative BTA injection on severity of surgical complications | During the 90-day postoperative period
  Severity of complications according to the Clavien-Dindo classification
Assessment of the impact of preoperative BTA injection on surgical difficulty: abdominal wall closure with CST; incomplete closure of the wall with need of bridge prosthetic repair | During IH repair surgery
  Occurrence of CST and occurrence of incomplete wall closure (bridge closure)
Assessment of the impact of preoperative BTA injection on radiological response:lateral muscles elongation | Between the pre-inclusion CT-scan and the CT-scan 4 weeks after BTA injection
  Sum of the length variation of the left and right lateral muscles (cm)
Assessment of the impact of preoperative BTA injection on radiological response:lateral muscles elongation | Between the pre-inclusion CT-scan and the CT-scan 4 weeks after BTA injection
  Sum of the width variation of the left and right lateral muscles (cm)
Assessment of the impact of preoperative BTA injection on radiological response: muscular defect reduction | Between the pre-inclusion CT-scan and the CT-scan 4 weeks after BTA injection
  Width (cm) variation of the muscular defect
Assessment of the impact of preoperative BTA injection on radiological response: muscular defect reduction | Between the pre-inclusion CT-scan and the CT-scan 4 weeks after BTA injection
  Surface(cm²) variation of the muscular defect
Assessment of the impact of preoperative BTA injection on radiological response: hernia sac volume | Between the pre-inclusion CT-scan and the CT-scan 4 weeks after BTA injection
  Volume (cm3) variation of the peritonial sac
Assessment of the impact of preoperative BTA injection on intra-abdominal pressure, monitored until bladder catheter removal | From catheter insertion to removal
  Measurement of intravesical pressure
Assessment of the impact of preoperative BTA injection on consequences of repair on pain evolution and consumption of analgesics | From 1st to 7th postoperative day and at 1, 3 , 6, and 12 months after surgery
  Pain on Analogical Visual Scale, prescription of type 3 analgesics
Assessment of the impact of preoperative BTA injection repair results: post-operative abdominal wall disruption , clinical and radiological recurrence of the IH | 90 days and 12 months after surgery
  Occurrence of post-operative abdominal wall disruption during a 90 days period after surgery, defined as early postoperative abdominal content herniation with or without skin coverage, identified clinically or at CT-scan; Occurrence of clinical recurrence of the IH during the first year after surgery, deﬁned as any fascial defect that was palpable and was located within 7 cm of the site of hernia repair while the patient was in the supine position with legs extended and raised.
  Occurrence of radiological recurrence of the IH at 12 months post-surgery; radiologic hernia is defined as any protrusion of abdominal contents including the anterior parietal peritoneum through a discontinuity of the fascial layers on CT performed during follow-up without Valsalva maneuver postoperative occurrence of clinical and radiological recurrence of the IH, or reoperation for recurrence.
Assessment of the impact of preoperative BTA injection on evolution of quality of life | 90 days, 6, and 12 months after surgery
  EQ-5D-5L scale

CONTACTS AND LOCATIONS:
Overall Officials: David MOSZKOWICZ, Principal Investigator — APHP
Locations (1):
- David Moszkowicz, Colombes, France, France

IPD SHARING:
Plan to Share IPD: No